CLINICAL TRIAL: NCT00703222
Title: A Phase I/II Study Of Immunization With Lymphotactin And Interleukin 2 Gene Modified Neuroblastoma Tumor Cells After High-Dose Chemotherapy And Autologous Stem Cell Rescue In Patients With High Risk Neuroblastoma
Brief Title: A Phase I/II Study Of Immunization With Lymphotactin And Interleukin 2 Gene Modified Neuroblastoma Tumor Cells
Acronym: CHESAT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Andras Heczey, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22053-CHESAT
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma
Keywords: high-risk neuroblastoma; single autologous stem cell rescue
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Intervention Model Description: Dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Dose Level 1 (Experimental): SNJB-JF-IL2 and SJNB-JF-Lptn + Dose Level 1 SKNLP
  Interventions: Biological: SNJB-JF-IL2 and SJNB-JF-Lptn + Dose Level 1 SKNLP
- Dose Level 2 (Experimental): SNJB-JF-IL2 and SJNB-JF-Lptn + Dose Level 2 SKNLP
  Interventions: Biological: SNJB-JF-IL2 and SJNB-JF-Lptn + Dose Level 2 SKNLP

INTERVENTIONS:
Biological: SNJB-JF-IL2 and SJNB-JF-Lptn + Dose Level 1 SKNLP — SJNB-JF-IL2 and SJNB-JF-Lptn at 1 x 10^7 cells/m2
  SKNLP at 1 x 10^6 cells/m2
  Arms: Dose Level 1
Biological: SNJB-JF-IL2 and SJNB-JF-Lptn + Dose Level 2 SKNLP — SJNB-JF-IL2 and SJNB-JF-Lptn at 1 x 10^7 cells/m2
  SKNLP at 1 x 10^7 cells/m2
  Arms: Dose Level 2

SUMMARY:
The investigators intend to test the safety, and immunologic and clinical efficacy of a combination of 2 allogeneic neuroblastoma tumor cell line vaccines, one of which has been genetically modified to secrete the cytokine/chemokine combination of IL-2 and lymphotactin, in patients undergoing chemotherapy for newly diagnosed, high risk neuroblastoma who receive single autologous stem cell rescue as consolidation therapy.

This protocol will be carried out as a Phase I/IIa study to evaluate the safety and toxicity of adding a previously unstudied, unmodified, irradiated neuroblastoma cell line (SKNLP) to a studied, safe dose of a gene modified, IL-2/Lptn secreting neuroblastoma cell line SJNB-JF-IL2/Lptn to be given as a vaccine to patients diagnosed with high risk neuroblastoma.

DETAILED DESCRIPTION:
TREATMENT PLAN: Standard Chemotherapy for Neuroblastoma: Standard therapy for neuroblastoma is given in 3 phases: induction, consolidation, and maintenance. For enrollment in this vaccine study patients and their physicians must anticipate therapy that will include consolidation with high dose chemotherapy with stem cell rescue. They will be eligible for enrollment in the phase I or phase II trial of vaccination with gene modified and unmodified, allogeneic neuroblastoma cell lines. Patients will receive Induction, Consolidation, and Maintenance therapy per their institutional standards. A general description of the therapy follows:

* Induction: Induction consists of multiple cycles of induction chemotherapy with harvest of autologous stem cells immediately following a particular cycle of chemotherapy per institutional standards. Local control of the tumor with radiation therapy and/or surgery occurs following a few cycles of induction chemotherapy or immediately prior to consolidation therapy.
* Consolidation: Consolidation must consist of high dose chemotherapy with autologous stem cell rescue (HDT/SCR).
* Maintenance: Starting day +90 after HDT/SCR, patients will be treated with Isotretinoin (Cis-Retinoic Acid, CRA).

VACCINE DOSING: Vaccine components SJNB-JF-IL2 and SJNB-JF-Lptn will each be dosed at 1x10e7 cells/m2. This will be given in conjunction with an escalating dose of SKNLP vaccine in the phase I portion of this study. In the phase II portion of this study, the same dose of SJNB-JF-IL2 and SJNB-JF-Lptn will be given in conjunction with the highest dose of SKNLP determined in the phase I portion. Vaccination will be administered on an inpatient or outpatient basis. Patient will be notified of which dose of vaccine cells they will receive if enrolled in the study.

Phase I Dose Escalation Component: While the investigators do not suspect that addition of a second irradiated, unmodified neuroblastoma tumor cell line to the previously tested SJNB-JF gene modified cell line will affect the safety profile of the vaccine, as the SKNLP has not been tested previously in vaccine studies, the investigators will perform an abbreviated dose escalation study of the combined vaccine to assess safety. The investigators know that the vaccine given to patients whose neuroblastoma returned was safe. The vaccine that was given to those patients was treated with the viruses to make cytokines. The investigators have never used the 2nd cell group in patients. Because of this, the investigators plan to treat 3 to 6 patients at a lower dose of cells to see if adding the second cell line is safe to give.

* Dose Level 1 (3-6 patients) 1x10e6 cells/m2/vaccination dose of SKNLP Unmodified Neuroblastoma Cell Line Vaccine Component
* Dose Level 2 (3-6 patients) 1x10e7 cells/m2/vaccination dose of SKNLP Unmodified Neuroblastoma Cell Line Vaccine Component

  * SJNB-JF-IL2 and SJNB-JF-Lptn cells are each dosed at 1x10e7 cells/m2/vaccination

Duration of Therapy: In the absence of treatment delays due to adverse events, treatment may continue with immunizations per the treatment plan up to 12 vaccinations or until one of the following criteria applies: - Disease progression - Intercurrent illness that prevents further administration of treatment - Unacceptable adverse events(s) including but not limited to grade 3-4 non-hematologic toxicity according to CTCAE v3.0. Grade 3 rigors/chills will be tolerated for 48-72 hours if attributed to vaccination. - Patient decides to withdraw from the study - General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgement of the investigator.

ELIGIBILITY:
Inclusion Criteria:

Age <21 years at time of diagnosis

Histological proof of high-risk neuroblastoma at diagnosis

Anticipating single autologous stem cell rescue following high dose consolidation chemotherapy

Meet all eligibility criteria for high dose chemotherapy with stem cell rescue per institutional standard

Signed informed consent

Patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. The male partner should use a condom.

HIV negative

Exclusion Criteria:

Patients must not be currently receiving any investigational agents or have received any tumor vaccines within the previous six months

Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Pregnant

HIV-positive patients regardless of treatment status

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-06; Primary Completion 2011-05 (Actual); Study Completion 2025-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of repeated immunization with gene-modified, IL-2/lymphotactin secreting SJNB-JF-IL2 and SJNB-JF-Lptn cells co-administered with the unmodified SKNLP neuroblastoma cell line. | 1 year
  21-day window following the first vaccination will constitute the time period for DLT assessment. Dose limiting toxicity will be any grade 3 or 4 non-hematologic toxicity as per the CTCAE v3.0 or a grade 3 injection site toxicity per the CTCAE 3.0. Toxicities after the initial as well as after subsequent vaccinations will be summarized separately.

SECONDARY OUTCOMES:
Evaluate the immune response to these immunizations. | 1 year
  Summarize ELISPOT levels of CTLp at baseline and each time point of assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Andras A. Heczey, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We will not share IPD with other researchers. Study outcomes will be published in aggregate.